CLINICAL TRIAL: NCT05074056
Title: Evaluation of Perioperative Usage of Ketorolac on Postoperative Pain Reduction in Pediatric Patients with Adenotonsillectom
Brief Title: Ketorolac on Postoperative Pain Reduction in Pediatric Patients with Adenotonsillectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Andrea Zepeda, MD, Associate Professor, SSM Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 31070
Record Dates: First submitted 2021-09-29; First posted 2021-10-12 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-09

CONDITIONS: Adenotonsillar Hypertrophy; Obstructive Sleep Apnea; Sleep-Disordered Breathing; Acute Post Operative Pain
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Pain, Postoperative | interventions — Ketorolac

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketorolac (Experimental): A double-blinded number of children will get one dose of intravenous 0.5 mg/kg (max dose 30mg) ketorolac intraoperatively.
  Interventions: Drug: Ketorolac
- Placebo (Placebo Comparator): A double-blinded number of children will get one dose of intravenous placebo intraoperatively.
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — We will administer intraoperative ketorlac.

SUMMARY:
Postoperative pain management in the pediatric patient undergoing tonsillectomy is challenging. Despite being used in many procedures for postoperative pain management, perioperative ketorolac usage in pediatric tonsillectomy surgery is very limited. A recent survey showed that only 8.2% of anesthesiologists use NSAIDS for perioperative management of children with OSA undergoing adenotonsillectomy. The investigators propose to conduct a prospective, randomized study to investigate the opioid-sparing effect of perioperative ketorolac in pediatric patients who undergo tonsillectomies.

DETAILED DESCRIPTION:
Adenotonsillectomy is one of the most frequent surgeries performed in pediatric population in the United States mainly due to conditions such as sleep disordered breathing and recurrent tonsillitis. However, postoperative pain control following adenotonsillectomy still offers great challenges to anesthesiologists. Postoperative pain has been the most common adverse effect in post-anesthesia care unit (PACU) for children undergoing tonsillectomies and postoperative pain is also correlated with emergence agitation, ileus, delayed mobilization, prolonged hospital stays, the development of chronic pain syndromes, and postoperative nausea and vomiting (PONV). Therefore, benefits of effective pain control are many fold: improving patient/family satisfaction, reducing the risk of postoperative bleeding due to emergence agitation, decreasing the incidence of PONV, and cutting down clinical symptoms related to opioid overdose.

To better control postoperative pain, pre-operative and intraoperative pain management have been the key. Preventative analgesic interventions may provide protection against the development of persistent postoperative pain. Although opioid derivatives such as fentanyl and morphine are mainstays for the perioperative management of post-tonsillectomy pain, opioid consumption is positively correlated with clinical adverse events such as PONV, opioid overdose, and over-sedation. Especially for pediatric patients with severe obstructive sleep apnea (OSA), opioids may depress ventilation and lead to further airway obstruction, resulting in desaturation of blood oxygen, and even death. Multi-modal pain control includes use of combinations of opioids with selective alpha2-adrenergic agonist such as dexmedetomidine and nonsteroidal anti-inflammatory drugs (NSAIDS) such as ketorolac, are frequently used for analgesia in children undergoing tonsillectomies. Dexmedetomidine is a selective alpha-2 adrenergic receptor agonist that directly acts on the peripheral nervous system, causing a dose-dependent inhibition of C-fibers and Aα-fibers. Non-selective NSAIDS have been shown to function both peripherally and centrally in nociception. NSAIDs act at the peripheral nociceptors by blocking the cyclooxygenase (COX) enzyme that inhibits the conversion of arachidonic acid to prostaglandins, thereby preventing the sensitization of pain receptors in response to injury. Centrally, NSAIDs inhibit prostaglandin E2 (PGE2) production in the spinal dorsal horn via COX-2, activate medullary and cortical brain regions involved in the descending inhibitory pain cascade, result in central sensitization and a lower pain threshold in the surrounding uninjured tissue.

Among NSAIDS, Ketorolac tromethamine (Toradol) is the first approved for parenteral use in 1990 in the United States. Despite its variety of clinical indications, it is mainly administered for the management of postoperative pain. It has strong analgesic properties, with a dose of 30 mg intramuscular (IM) offering similar analgesia as 12 mg of morphine. The strong analgesic properties of reducing opioid requirements make it a good candidate in multi-modal pain management of post-tonsillectomy pain. Unlike opioid analgesics, ketorolac does not depress ventilation, and is not associated with nausea and vomiting, urinary retention or sedation. When combined with an opioid, ketorolac exhibits significant opioid-sparing effects, allowing a lower dosage of opioid to be used. Clinical studies in children and adults show that the synergistic action of ketorolac and opioids improves the degree and quality of pain relief, and reduces the incidence of opioid-related adverse effects such as respiratory depression, PONV, and ileus. However, similar to other non-selective Cox enzyme inhibitors, ketorolac has several adverse effects including gastrointestinal (GI) bleeding, renal impairment, liver dysfunction, possible allergic reactions, and disruption of platelet aggregation through the inhibition of thromboxane A. However, the evidence of increased bleeding is conflicting. A meta-analysis suggested that there was no consensus on the increased risk of bleeding when NSAIDS such as ketorolac are given to pediatric patients undergoing tonsillectomy. There are other analyses to support that conclusion.

Despite of these findings, perioperative ketorolac usage, especially in pediatric tonsillectomy surgery, is very limited.

ELIGIBILITY:
Inclusion Criteria:

* Adenotonsillar hypertrophy
* ASA II
* Otherwise healthy child

Exclusion Criteria:

* Child < 3 years old and > 12 years old
* Severe Obstructive sleep apnea
* Chronic Kidney disease
* Chronic Liver Disease

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 142 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Postoperative pain management | two hours
  Change in pain score using the Wong-Baker FACES Pain Rating Scale (0-10 scale with 0 being "no hurt" and 10 being "hurts worst") and 0-10 Numeric Pain Intensity Scale (0-10 scale with 0 being "no pain" and 10 being "Worst pain").

CONTACTS AND LOCATIONS:
Locations (1):
- SSM Cardinal Glennon Children's Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Franz AM, Dahl JP, Huang H, Verma ST, Martin LD, Martin LD, Low DK. The development of an opioid sparing anesthesia protocol for pediatric ambulatory tonsillectomy and adenotonsillectomy surgery-A quality improvement project. Paediatr Anaesth. 2019 Jul;29(7):682-689. doi: 10.1111/pan.13662. Epub 2019 Jun 19. PMID 31077491
- [Background] Tan GX, Tunkel DE. Control of Pain After Tonsillectomy in Children: A Review. JAMA Otolaryngol Head Neck Surg. 2017 Sep 1;143(9):937-942. doi: 10.1001/jamaoto.2017.0845. PMID 28662233
- [Background] Scalzitti NJ, Sarber KM. Diagnosis and perioperative management in pediatric sleep-disordered breathing. Paediatr Anaesth. 2018 Nov;28(11):940-946. doi: 10.1111/pan.13506. Epub 2018 Oct 3. PMID 30281185
- [Background] Tang C, Xia Z. Dexmedetomidine in perioperative acute pain management: a non-opioid adjuvant analgesic. J Pain Res. 2017 Aug 11;10:1899-1904. doi: 10.2147/JPR.S139387. eCollection 2017. PMID 28860845
- [Background] Gupta A, Bah M. NSAIDs in the Treatment of Postoperative Pain. Curr Pain Headache Rep. 2016 Nov;20(11):62. doi: 10.1007/s11916-016-0591-7. PMID 27841015
- [Background] Cashman JN. The mechanisms of action of NSAIDs in analgesia. Drugs. 1996;52 Suppl 5:13-23. doi: 10.2165/00003495-199600525-00004. PMID 8922554
- [Background] Vadivelu N, Chang D, Helander EM, Bordelon GJ, Kai A, Kaye AD, Hsu D, Bang D, Julka I. Ketorolac, Oxymorphone, Tapentadol, and Tramadol: A Comprehensive Review. Anesthesiol Clin. 2017 Jun;35(2):e1-e20. doi: 10.1016/j.anclin.2017.01.001. Epub 2017 Apr 14. PMID 28526155
- [Background] Maslin B, Lipana L, Roth B, Kodumudi G, Vadivelu N. Safety Considerations in the Use of Ketorolac for Postoperative Pain. Curr Drug Saf. 2017;12(1):67-73. doi: 10.2174/1574886311666160719154420. PMID 27440142
- [Background] Forrest JB, Heitlinger EL, Revell S. Ketorolac for postoperative pain management in children. Drug Saf. 1997 May;16(5):309-29. doi: 10.2165/00002018-199716050-00003. PMID 9187531
- [Background] Forrest JB, Camu F, Greer IA, Kehlet H, Abdalla M, Bonnet F, Ebrahim S, Escolar G, Jage J, Pocock S, Velo G, Langman MJ, Bianchi PG, Samama MM, Heitlinger E; POINT Investigators. Ketorolac, diclofenac, and ketoprofen are equally safe for pain relief after major surgery. Br J Anaesth. 2002 Feb;88(2):227-33. doi: 10.1093/bja/88.2.227. PMID 11883386
- [Background] Phillips-Reed LD, Austin PN, Rodriguez RE. Pediatric Tonsillectomy and Ketorolac. J Perianesth Nurs. 2016 Dec;31(6):485-494. doi: 10.1016/j.jopan.2015.02.005. Epub 2016 May 5. PMID 27931700
- [Background] Lewis SR, Nicholson A, Cardwell ME, Siviter G, Smith AF. Nonsteroidal anti-inflammatory drugs and perioperative bleeding in paediatric tonsillectomy. Cochrane Database Syst Rev. 2013 Jul 18;2013(7):CD003591. doi: 10.1002/14651858.CD003591.pub3. PMID 23881651
- [Background] Roberts C, Al Sayegh R, Ellison PR, Sedeek K, Carr MM. How Pediatric Anesthesiologists Manage Children with OSA Undergoing Tonsillectomy. Ann Otol Rhinol Laryngol. 2020 Jan;129(1):55-62. doi: 10.1177/0003489419874371. Epub 2019 Sep 5. PMID 31801377